CLINICAL TRIAL: NCT04090606
Title: Constituent Yields and Biomarkers of Exposure for Tobacco Product Regulation
Brief Title: Tobacco Constituents and Biomarkers
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2013NTLS115
Record Dates: First submitted 2019-09-10; First posted 2019-09-16 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FTC Method
  Interventions: Other: FTC Method Smoking Regimen
- Massachusetts Method
  Interventions: Other: Massachusetts Method Smoking Regimen
- Health Canada Intense Method
  Interventions: Other: Health Canada Intense Smoking Regimen

INTERVENTIONS:
Other: FTC Method Smoking Regimen — cigarettes are smoked by drawing 35 mL puff volumes over 2 s, with 60 s interval between puffs and no blocking of filter ventilation holes
  Groups: FTC Method
Other: Massachusetts Method Smoking Regimen — 45-mL puffs drawn over 2 s, with 30 s interval between puffs and 50% blocking of filter ventilation holes
  Groups: Massachusetts Method
Other: Health Canada Intense Smoking Regimen — 55-mL puff volumes of 2-s duration, with 30 s interval between puffs and 100% blocking of filter ventilation holes
  Groups: Health Canada Intense Method

SUMMARY:
This proposal addresses several research priorities related to the regulatory authority of the Food and Drug Administration (FDA) Center for Tobacco Products as mandated by the Family Smoking Prevention and Tobacco Control Act. Scientific evidence supports the important role of tobacco and cigarette smoke carcinogens in the development of cancers associated with cigarette smoking. Regulation of the levels of harmful constituents in cigarette smoke is one of the tobacco control strategies that now can be employed by the FDA and may serve to reduce tobacco carcinogen exposures in those smokers who are unable or unwilling to quit smoking. Such regulation will require a valid and robust approach to the assessment of comparative toxicity and carcinogenicity among various cigarette brands. This proposal will help develop a testing approach that can produce meaningful predictions of changes in human exposure due to changes in constituent levels in cigarette smoke, and hence serve as a reliable measure for product regulation. Thus, the proposed research will generate findings and data that are directly relevant to inform the FDA's regulation of the manufacture, distribution, and marketing of tobacco products to protect public health. The human trial deals with Aims 2 and 3 of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult smokers 18-65 years of age, who smoke at least 7 cigarettes per day (to assure that biomarker levels are above the limit of quantitation) and do not have plans to quit smoking in the next month;
* Smoked the same brand for >80% of their cigarettes over the course of at least 1 year, and smoked not more than 20 cigarettes (1 pack) of a different brand within two weeks prior to the eligibility screening;
* Not using any other nicotine or tobacco product;
* Subjects who are not taking any medications that affect relevant metabolic enzymes;
* Women who are not pregnant or nursing;
* Subjects have provided written informed consent to participate in the study (adolescents under the age of 18 will be excluded because this project involves use of tobacco products).

Exclusion Criteria:

* Significant immune system disorders, respiratory diseases, kidney or liver diseases or any other medical disorders that may affect biomarker data;
* Current or recent alcohol or drug abuse problems (to ensure alcohol and drug use does not affect biomarkers of exposure and to maximize retention);
* Regular tobacco use (e.g., greater than weekly) other than cigarettes;
* Currently using nicotine replacement or other tobacco cessation products (to minimize confounding effects of another product);
* Pregnant or breastfeeding (due to toxic effects from tobacco products)
* Report smoking more than 1 pack (20 cigarettes) of a non-usual brand cigarette in the past two weeks * Participants who report smoking 2 or more non-usual brand cigarettes the day before the clinic visit will be ineligible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult smokers from Minneapolis-St. Paul metro area
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
The extent to which differences in smoke yields of NNN and NNK per mg nicotine are predictive of differences in smokers' exposure to these carcinogens (human trial) | 1 Year
  Correlation between urinary total NNN and total NNAL (with and without normalization for total nicotine intake) in smokers and the machine-measured yields of NNN and NNK (per mg nicotine and per cigarette) in cigarettes smoked by these individuals. The relationship will be investigated for the machine-measured yields generated by 3 different smoking regimens.
The extent to which NNN and NNK per mg nicotine levels in spent cigarette filters are predictive of differences in smokers' exposure to these carcinogens (human trial) | 1 Year
  Correlation, for each smoker, between the TSNA per mg nicotine content in their spent cigarette filters with the levels of total NNN and total NNAL per nicotine equivalents in their urine

SECONDARY OUTCOMES:
Individual factors affecting TSNA per mg nicotine and exposures in smokers (human trial) | 1 Year
  Correlation (if any) of individual factors and the relationship between the machine-measured TSNA per mg nicotine and exposures in smokers.
Relationship between 1-HOP and TSNA per mg Nicotine | 1 Year
  Correlation between urinary biomarker of polycyclic aromatic hydrocarbon exposure (1-HOP) and TSNA per mg nicotine yields in cigarette smoke.